CLINICAL TRIAL: NCT07031947
Title: The Effect of Core Stabilization Exercise Program Applied With Telerehabilitation Method in Virtual Reality Environment in the Treatment of Patients With Chronic Non-Specific Low Back Pain: A Single-Blind Randomized Controlled Study
Brief Title: The Effect of Core Stabilization Exercises Applied With Virtual Reality-Based Telerehabilitation in the Treatment of Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Istanbul University Research Fund (Unknown)
Responsible Party: Principal Investigator, Emre Öney, Medical Doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-29624016-050.04-2603725
Record Dates: First submitted 2025-06-01; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain; Low Back Pain, Mechanical; Low Back Pain and Core Muscle; Core Stabilization Exercise Therapy
MeSH Terms: conditions — Low Back Pain | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (Active Comparator)
  Interventions: Other: Core stabilization exercise with telerehabilitation
- Face-to-face rehabilitation group (Other)
  Interventions: Other: Face-to-face core stabilization exercise

INTERVENTIONS:
Other: Core stabilization exercise with telerehabilitation — In addition to a brochure containing patient education, showing the application method of core stabilization exercises, the number of sets and repetitions, the intervention group (G1) will receive a back school program in a total of 2 sessions of videoconference interviews, and the exercises will be explained to them, supported by visuals and videos. In addition, patients will be provided with the application that will be provided with your support, and will be provided with core stabilization exercises 3 times a week for 8 weeks.
  Arms: Telerehabilitation Group
Other: Face-to-face core stabilization exercise — The control group (G2) will receive a brochure that includes patient education, showing the application method of core stabilization exercises, the number of sets and repetitions, as well as a face-to-face back school program in our hospital for a total of 2 sessions. The exercise program will be carried out face to face, 3 sessions per week for 8 weeks, at the Istanbul University, Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, under the supervision of a physician, with each exercise session being in groups of 8 people.
  Arms: Face-to-face rehabilitation group

SUMMARY:
A total of 80 patients, aged between 20 and 60 years, diagnosed with non-specific low back pain and not meeting the exclusion criteria, who registered at the outpatient clinics of the Department of Physical Medicine and Rehabilitation, Istanbul University, Istanbul Faculty of Medicine, between June 1, 2024 and June 1, 2025, were planned to be included in our thesis study, which was planned to be prospective, randomized and single-blind. After the patients are informed verbally and in writing about the purpose, duration and application method of the study and their consent is obtained, they will be asked to sign the "Informed Consent Form". Patient evaluation and follow-up forms will be filled out during pre-treatment and post-treatment follow-ups. After patients who meet the study inclusion criteria are included in the study, they will be numbered according to the order of application and then randomly assigned to the intervention group or control group by a computer program into 2 groups.

In addition to a brochure containing patient education, showing the application method of core stabilization exercises, the number of sets and repetitions, the intervention group (G1) will receive a back school program in a total of 2 sessions of videoconference interviews, and the exercises will be explained to them, supported by visuals and videos. In addition, patients will be provided with the application that will be provided with your support, and will be provided with core stabilization exercises 3 times a week for 8 weeks.

The control group (G2) will receive a brochure that includes patient education, showing the application method of core stabilization exercises, the number of sets and repetitions, as well as a face-to-face back school program in our hospital for a total of 2 sessions. The exercise program will be carried out face to face, 3 sessions per week for 8 weeks, at the Istanbul University, Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, under the supervision of a physician, with each exercise session being in groups of 8 people.

ELIGIBILITY:
Inclusion Criteria:

Between 20 and 60 years of age Non-specific low back pain lasting more than 3 months (VAS > 2) No neurological deficits such as abnormal sensation, loss of muscle strength, or loss of reflexes in the lower extremity No indication for surgery Able to attend treatment 3 days a week for 8 weeks

Exclusion Criteria:

Participating in a physical therapy or exercise program in the last 3 months Previous surgery, dislocation, or fracture in the lumbar region Rheumatic / autoimmune disease Serious cardiovascular disease, progressive neurological deficit, severe osteoporosis, or metabolic diseases Having a systemic disease that can cause back pain Pregnancy or lactation Uncontrolled hypertension Having problems perceiving verbal commands Not having internet access Not having equipment to make video calls at home Not having a device at home to use the application

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Oswestry Low Back Pain Disability Index | Day 1 (before starting treatment), Day 60 (end of treatment), Day 120 (two months after the end of treatment)
  It is a commonly used and validated scale for measuring disability in low back pain. It consists of a total of 10 questions. Each question is scored on a scale of 0 to 5. Higher scores indicate worse symptoms or functioning.
Visuel Analog Scale | Day 1 (before starting treatment), Day 60 (end of treatment), Day 120 (two months after the end of treatment)
  The severity of pain before treatment is assessed using the Visual Analog Scale (VAS), a 10 cm long line with "no pain" on the left end and "unbearable pain" on the right end. The distance in centimeters between the point marked by the patient and the 0 point is measured. The average pain level before and after treatment will be evaluated using the VAS, scored between 0 and 10; 0 indicates no pain, and 10 indicates the worst possible pain.

SECONDARY OUTCOMES:
Roland Morris Disability Questionnaire | Day 1 (before starting treatment), Day 60 (end of treatment), Day 120 (two months after the end of treatment)
  It is a validated scale used to measure disability in low back pain. The total score ranges from 0 (no disability) to 24 (severe disability). A higher total score indicates decreased patient functionality. Higher scores reflect worse symptoms or function.
Tampa Kinesiophobia Fatigue Scale | Day 1 (before starting treatment), Day 60 (end of treatment), Day 120 (two months after the end of treatment)
  The Tampa Scale for Kinesiophobia is a 17-item tool used to assess fear of movement. A 4-point Likert scoring system is used in the questionnaire. Items 4, 8, 12, and 16 are reverse scored, and the total score is calculated by summing all items. The total score ranges from 17 to 68. A higher score on the scale indicates a higher level of kinesiophobia.
Measurement of Bilateral Lumbar Multifidus and Transversus Abdominis Muscle Thickness with Ultrasound Imaging | Day 1 (before starting treatment), Day 60 (end of treatment), Day 120 (two months after the end of treatment)
  Ultrasonographic evaluation will be performed using the Esaote Mylab 60 device. The resting muscle thickness of the lumbar multifidus will be measured longitudinally with a convex probe at the L4-L5 facet level at the end of expiration while the patient is in the prone position. After the contralateral arm-raising maneuver, the contracted thickness of the multifidus will be measured at the same level.
  The transversus abdominis measurement will be performed at the end of expiration in the supine position, with knees bent, heels resting on the table, and hands placed under the head. A linear probe will be used at the midpoint between the 12th rib and the iliac crest, 2.5 cm anterior to the mid-axillary line. Following the ipsilateral straight leg raise maneuver, the contracted transversus abdominis thickness will be measured at the same level.
Assessment of Trunk Muscle Strength with Computerized Isokinetic Dynamometer | Day 1 (before starting treatment), Day 60 (end of treatment), Day 120 (two months after the end of treatment)
  In our study, trunk extensor and flexor muscle strengths will be measured with a Biodex System 3-Pro (Biodex Medical Systems, Inc, New York, USA) computerized isokinetic dynamometer machine. Maximum strength will be used to perform trunk extension and flexion at speeds of 60°/s, 90°/s, and 120°/s, respectively, with 5 repetitions at each speed. Peak torque and total work values of the participants will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Unıversity, Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided